CLINICAL TRIAL: NCT06777121
Title: Effects of Adding Thoracic Extension Exercises or Thoracic Kinesio Taping to Shoulder Exercises on Pain, Function, Range of Motion, Strength, and Thoracic Kyphosis in Adults With Subacromial Pain Syndrome
Brief Title: Effects of Exercise or Taping on Pain, Function, Range of Motion, Strength and Kyphosis in Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevtap Günay (Other)
Responsible Party: Sponsor-Investigator, Sevtap Günay, Associate Professor, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KatipCelebiUniversity
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Subacromial Impingement Syndrome; Exercise Addiction; Shoulder Pain
Keywords: Shoulder pain; Shoulder function; Shoulder exercise; Kinesio taping; Thoracic exercise; Thoracic posture
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: This research was planned as a randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The evaluator did not know the group to which the participants were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): In addition to shoulder exercises, thoracic extension exercises were performed.
  Interventions: Other: Shoulder exercises + Thoracic extension exercise
- Group B (Active Comparator): In addition to shoulder exercises, kinesio taping was applied.
  Interventions: Other: Shoulder exercises + Thoracic kinesio taping
- Group C (Active Comparator): Only shoulder exercises were performed.
  Interventions: Other: Shoulder exercises

INTERVENTIONS:
Other: Shoulder exercises + Thoracic extension exercise — Shoulder exercises and thoracic extension exercises were performed 5 days a week for 3 weeks.
  Arms: Group A
Other: Shoulder exercises + Thoracic kinesio taping — In addition to shoulder exercises, thoracic kinesio taping was applied. Shoulder exercises were performed 5 days a week for 3 weeks. TKT was applied once a week and remained in place for 5 days.
  Arms: Group B
Other: Shoulder exercises — Shoulder exercises were performed. They were performed 5 days a week for 3 weeks.
  Arms: Group C

SUMMARY:
Participants with subacromial pain syndrome underwent shoulder exercises. In addition to the exercises, group A received thoracic extension exercise and group B received kinesio taping. All exercises were performed five days per week for three weeks. Thoracic extension exercise was performed once a week and remained in place for 5 days. Evaluations were performed one to three days before and one to three days after the three-week exercise program.

DETAILED DESCRIPTION:
Seventy-five adults with subacromial pain syndrome were randomized into three groups. Group A and Group B received thoracal extension exersice and thoracal kinesiotaping in addition to shoulder exercise, respectively, while Group C received only shoulder exercise. All exercises were performed five days a week for three weeks. Thoracal extension exercise was applied once a week and remained in place for 5 days. Assessments were conducted one to three days before and one to three days after the three-week exercise program. Shoulder pain intensity, pressure pain threshold (PPT) of the upper trapezius and pectoralis major, self-reported function and health status, active range of motion (AROM), and isometric strength of the shoulder were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Having shoulder pain for at least 6 weeks
* Aggravation of shoulder pain with resisted shoulder movements

Exclusion Criteria:

* Those with full-thickness rotator cuff rupture
* Those who have had previous shoulder surgery
* Those who have had cervical or thoracic spine surgery
* Those with a history of inflammatory disease or cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Shoulder function assessment | At the beginning and after 3 weeks
  Disabilities of the Arm, Shoulder and Hand Questionnaire was used to assess the condition. It is a questionnaire used to evaluate upper extremity function status. The questionnaire consists of three sections, and the person marks the appropriate answer for each question on the Likert system with a score of 5 (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: completely unable to do). According to the DASH questionnaire result; a result between 0-100 is obtained from each section.
Muscle strength assessment | At the beginning and after 3 weeks
  Muscle strength will be measured with a digital hand dynamometer. Muscle strength measurements of the subjects' flexion, extension abduction, adduction, external and internal rotation movements will be made. The measurements made with the dynamometer will be based on the fine muscle test positions and method defined by Lovett. The tests will be repeated three times and at least one minute of rest will be given between repetitions. The highest of the 3 repetitions was accepted as the result.
Thoracic kyphosis assessment | At the beginning and after 3 weeks
  For thoracic kyphosis measurement, inclinometers were placed at T1-T2 and T12-L1 to perform the evaluation.
Pain intensity assessment | At the beginning and after 3 weeks
  It was evaluated using a visual analog scale. The scale is between 0 and 10 points, and increasing numbers indicate increased pain intensity.
Pressure pain threshold assessment | At the beginning and after 3 weeks
  Pressure pain threshold measurement was measured with an algometer device. Algometers are a device that can be used to define pressure and pressure pain threshold. Upper trapezius and pectoralis major muscles were evaluated.
Quality of life assessment | At the beginning and after 3 weeks
  Health-related quality of life (SF-36) was assessed with the questionnaire. It consists of 36 items in total and has eight sub-parameters. These eight sub-parameters consist of physical function, pain, social function, physical role limitations, mental health, emotional role limitations, vitality, and general health parameters. The sub-scales are scored between 0-100 and an increase of 26 points indicates an increase in the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap GUNAY UCURUM, Assoc. Dr., Principal Investigator — Izmir Katip Çelebi University, Department of Physiotherapy and Rehabilitation; Müge KIRMIZI, dr. lecturer, Principal Investigator — Izmir Katip Çelebi University, Department of Physiotherapy and Rehabilitation; Ayşenur YUKSEL, PT, Study Chair — Department of Physiotherapy and Rehabilitation, Bakircay University Training and Research Hospital
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No